CLINICAL TRIAL: NCT05344443
Title: Effect of a Dual Orexin Receptor Antagonist, Lemborexant, on Total Sleep Time in Shift Workers: a Randomized Controlled Trial
Brief Title: Lemborexant Shift Work Treatment Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-32763
Record Dates: First submitted 2022-03-10; First posted 2022-04-25 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Shift-Work Related Sleep Disturbance
Keywords: Shift Work; Daytime Sleepiness; Lemborexant
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: This will be a 4-week double blinded placebo controlled trial (2 weeks of baseline assessment followed by 2-weeks of treatment/placebo). The trial design is based on a recent successful study of the treatment of sleep problems in shift workers with a hypocretin/orexin receptor antagonist
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment (Experimental): Participants randomized into this arm will receive Lemborexant (5-10mg).
  Interventions: Drug: Lemborexant
- Placebo Treatment (Placebo Comparator): Participants randomized into this arm will receive a placebo medication which appears the same as the active treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant — A dual orexin antagonist
  Other Names: Dayvigo
  Arms: Active Treatment
Drug: Placebo — A placebo that looks and tastes like Lemborexant tablets
  Arms: Placebo Treatment

SUMMARY:
Insomnia and daytime sleepiness are common complaints among night shift workers, but effective sleep treatments in shift workers are lacking. The aim of this Phase IV double-blind, placebo-controlled, randomized study is to test whether a dual orexin antagonist, Lemborexant (5mg or 10mg), which would be expected to block the clock-driven orexin-mediated wakefulness during the day, will increase daytime sleep time in shift workers who complain of difficulty sleeping during the daytime compared to placebo.

DETAILED DESCRIPTION:
Insomnia and daytime sleepiness are common complaints among night shift workers. A meta-analysis on sleep in shift workers indicates that fixed night shift workers sleep, on average, 0.4 hours less than fixed day shift workers, while rotating shift workers sleep on average 1 hour less than fixed day shift workers. While there may be several reasons for sleep difficulties and sleep loss among shift workers, the misalignment of one's sleep preference (i.e., goal of sleeping during the day) and one's circadian rhythm (i.e., endogenous rhythm that signals the body to be awake during the day) is thought to be a primary cause. Insufficient sleep among night shift and rotating shift workers is linked with significant health consequences, including elevated risk for cardiovascular disease and cancer. Effective sleep treatments in shift workers are lacking. However, a recent randomized study of Suvorexant (20mg), a hypocretin/orexin receptor antagonist, produced a significant improvement in daytime total sleep time compared to placebo. Available evidence suggests that the reason Suvorexant is effective is because it blocks the hypocretin/orexin receptors that mediate signaling from the biological clock (suprachiasmatic nucleus of the hypothalamus) attempting to maintain sustained wakefulness during the biological day. As Lemborexant is also a hypocretin/orexin antagonist, it would also be expected to improve daytime sleep in shift workers but would have the advantage over Suvorexant of being highly effective in the dosages available for clinical use. As such, Lemborexant is ideally positioned to be an effective and important treatment of sleep problems in shift workers.

The aim of this Phase IV double-blind, placebo-controlled, randomized study is to test whether a dual orexin antagonist, Lemborexant (5mg or 10mg), which would be expected to block the clock-driven orexin-mediated wakefulness during the day, will increase daytime sleep time in shift workers who complain of difficulty sleeping during the daytime compared to placebo.

This will be a 4-week double blinded placebo controlled trial (2 weeks of baseline assessment followed by 2-weeks of treatment/placebo). The trial design is based on a recent successful study of the treatment of sleep problems in shift workers with a hypocretin/orexin receptor antagonist.

ELIGIBILITY:
Inclusion Criteria:

* Full-time night shift work (at least 6 hours per shift, 4 days per week or 32 hours per week)
* Employed as a night shift worker for at least 3 months
* Self-reported concerns about daytime sleepiness and difficulty sleeping during the daytime

Exclusion Criteria:

* Pregnancy (verified by urine pregnancy test) or plan to become pregnant in the next 3 months
* Currently breastfeeding
* Inadequate opportunity for sleep during the daytime (< 7 hours opportunity) after overnight shift
* Extreme circadian preference (based on Horne & Ostberg Morningness-Eveningness Questionnaire)
* Severe depressive symptoms (>25 on CES-D)
* Unwillingness to discontinue sleep aids (prescription or non-prescription) during the study period
* Presence of sleep disordered breathing (verified by Apnea link)
* Self-reported diagnosis of narcolepsy, restless legs syndrome
* Self-reported intake of >600mg of caffeine per night shift or use of stimulants during night shift, rotational, or irregular shifts
* Unstable or untreated medical or psychiatric condition based on clinical interview.
* Severe hepatic or renal impairment (based on chemistry panel);
* Self-reported use of digoxin or strong or moderate cytochrome P450 3A4 isozyme inhibitors or cytochrome P450 3A4 isozyme inducers for 6 months prior to or during the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aric Prather, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Screener — http://tinyurl.com/UCSFShiftStudy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants began in March 2022 and ended in December 2024. Participants were recruited primarily through flyers, with targeted recruitment at local hospitals.
Pre-assignment Details: Study participants completed baseline assessments, including sociodemographic questionnaires, clinical labs, and sleep measures (diaries, actigraphy) prior to randomization.
Period: Overall Study
Arm/Group | Active Treatment | Placebo Treatment
Started | 15 | 14
Completed | 15 | 13
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] — Self-reported age as a continuous measure in years Population: 1 participant in the active treatment group did not provide their age.
  Years
    number analyzed (Participants) | 14 | 14 | 28
    (all) | 37.8 (9.3) | 36.6 (8.4) | 37.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported biological sex
  Participants
    Female | 15 | 13 | 28
    Male | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported race/ethnicity
  Participants
    White/Caucasian | 4 | 8 | 12
    Black/African American | 2 | 1 | 3
    Asian | 7 | 2 | 9
    Hispanic/Latino | 2 | 2 | 4
    Multiracial | 0 | 1 | 1
Region of Enrollment [Number; unit: Participants] — Location
  Participants
    United States | 15 | 14 | 29
Diary-based daytime total sleep time [Mean (Standard Deviation); unit: Minutes per day] — Daytime total sleep time in minutes per day following a night shift averaged over the two-week baseline period Population: Two participants in the active treatment and two participants in the placebo group were missing diary based total sleep time value at baseline.
  Minutes per day
    number analyzed (Participants) | 13 | 12 | 25
    (all) | 341.1 (78.9) | 332.9 (66.2) | 336.8 (71.2)
Actigraphy-based daytime total sleep time [Mean (Standard Deviation); unit: Minutes per day] — Actigraphy daytime total sleep time in minutes per day following a night shift averaged over the two-week baseline Population: Six participants in the active treatment and 5 participants in the placebo condition were missing usable actigraphy data at baseline.
  Minutes per day
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 322.6 (125.2) | 286.4 (59.8) | 304.5 (97.0)

OUTCOME MEASURES:

1. Primary Outcome: Daytime Total Sleep Time in Minutes Per Day Collected From the Consensus Sleep Diary
Description: Daytime total sleep time in minutes per day following a night shift averaged over the two-week treatment/placebo period. Daytime total sleep time in minutes per day was recorded using the Consensus Sleep Diary, which participants completed daily.
Time Frame: Two weeks of Treatment
Population: Sleep diaries completed during daytime sleep attempts were the source of the treatment data. However, one participant (in the drug condition) failed to provide any useable diaries for daytime sleep attempts
Measure: Mean (Standard Error); unit: Minutes per day
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 14 | 14
Minutes per day | 362.7 (22.0) | 365.3 (22.4)
Statistical Analysis 1: Comparison: Active Treatment vs Placebo Treatment; We carried out linear mixed models to test the effect of condition on change in daytime sleep minutes from baseline to post-treatment. This analysis was powered based on prior literature (Zeitzer et al., 2020), which detected an effect size (Cohen's d) of 1.39 in a sample size of 19 participants; Test type: Superiority; p = 0.884, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05; Mean Difference (Net) = -5.9, 95% CI 2-sided [-88.3 to 76.4] — This linear mixed model included condition, time, and condition*time as fixed effect and a random intercept. It included "number of entries" as a random effect due to the fact that participants differed in number of diaries contributing to data

2. Secondary Outcome: Daytime Total Sleep Time in Minutes Per Day Measured by Actigraphy
Description: Daytime total sleep time in minutes per day following a night shift averaged over the two-week treatment/placebo period. Daytime total sleep time in minutes per day was collected using daily actigraphy data from Actiwatches, which participants wore during the two week treatment period.
Time Frame: Two weeks of treatment
Population: These analyses rely on wrist actigraphy data collected post-treatment. No actigraphy data were available in In 3 participants randomized to the placebo group and 1 participant in the drug condition.
Measure: Mean (Standard Error); unit: Minutes per day
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 14 | 11
Minutes per day | 318.4 (21.1) | 324.0 (29.2)
Statistical Analysis 1: Comparison: Active Treatment vs Placebo Treatment; Test type: Superiority; p = 0.494, Mixed Models Analysis; P-values were obtained from a linear mixed-effects model using restricted maximum likelihood estimation. Includes random intercept; Mean Difference (Net) = -40.2, 95% CI 2-sided [-159.2 to 78.7] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Events were collected beginning at randomization until the end of follow-up, up to 5 weeks.
Description: Adverse events were assessed by an open-ended question by the PI. Details on the event, the duration, and the likelihood of whether the event was related to study medication was obtained.
Arm/Group | Active Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 5/15 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=15) | Placebo Treatment (N=14)
Grogginess (General disorders) | 4 (5) | 0 (0)
Vivid dreaming/nightmare (General disorders) | 3 (3) | 0
Fragmented sleep (General disorders) | 3 (4) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1)
Sleep paralysis (General disorders) | 2 (2) | 0
Twisted ankle (General disorders) | 1 (1) | 0 (0)
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to challenges in recruitment and difficulties obtaining daytime sleep diaries and wrist actigraphy data, this study is likely underpowered, and the findings should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT05344443/Prot_SAP_000.pdf